CLINICAL TRIAL: NCT06780540
Title: Testing and Evaluating a Psychoeducational Toolkit and Clinical Screening Guidelines for Victims of Domestic and Sexual Violence in Belgian Hospitals.
Brief Title: Testing and Evaluating a Psychoeducation Tool and Guidelines for Victims of Violence in Belgian Hospitals.
Acronym: Operatie Alert
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Delta (Other); Centre Hospitalier Universitaire de Liege (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Vertrouwenscentrum Kindermishandeling (Unknown); Aditi ASBL/vzw (Unknown); SOS enfants asbl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ONZ-2024-0077; PSY/JO/Programma IFG-SG-VGV/20 (Other Grant/Funding Number: FOD Volksgezondheid)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Enhance Care to Victims of Violence
Keywords: violence; abuse; psycho-education; guideline; training; pilot study; clinical trial; evaluation; Belgium; hospitals; victims; healthcare providers; mixed methods research; multi-method design; sexual violence; domestic violence; older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operation Alert: Support program (Experimental): Substudy 1:
  Testing of a newly developed psycho-education tool will occur across four partner hospitals and participating nonprofit organizations (NGOs). Victims of violence seeking care at these sites will receive immediate support, with the pilot study integrated into standard care practices. The psycho-education toolkit enhances the foundational care already provided. The tool supports healthcare providers in offering psycho-education about e.g. violence and (the effects) of trauma, ...
  Substudy 2:
  This pilot study evaluates the Operation Alert guidelines within the geriatrics departments of four hospitals. A geriatric assessment is standard care during admission to these departments. The pilot will be embedded into this existing practice to ensure alignment with routine care. Additional questions will be embedded in a geriatric assessment/intake focusing on older adults' well-being, relationships and social network, and potential life events (e.g. experiences of violence).
  Interventions: Other: Operation Alert: Support prgram

INTERVENTIONS:
Other: Operation Alert: Support prgram — Substudy 1:
  Testing of a newly developed psycho-education tool will occur across four partner hospitals and participating nonprofit organizations (NGOs). Victims of violence seeking care at these sites will receive immediate support, with the pilot study integrated into standard care practices. The psycho-education toolkit enhances the foundational care already provided. The tool supports healthcare providers in offering psycho-education about e.g. violence and (the effects) of trauma, ...
  Substudy 2:
  This pilot study evaluates the Operation Alert guidelines within the geriatrics departments of four hospitals. A geriatric assessment is standard care during admission to these departments. The pilot will be embedded into this existing practice to ensure alignment with routine care. Additional questions will be embedded in a geriatric assessment/intake focusing on older adults' well-being, relationships and social network, and potential life events (e.g. experiences of violence).

SUMMARY:
The "Operation Alert/Operatie Alert/Opération Alerte" project, developed by UGent-ICRH and UZGent with funding from the Belgian Federal Public Service for Health, focuses on strengthening basic competencies to better and more quickly identify signs of violence. It also aims to provide victim-centered care and refer to specialized services when necessary. This initiative combines training for healthcare providers with practical tools, such as a psycho-education tool and clinical guidelines, to enhance care delivery. Below is an overview of the project's main components:

Sub-Study 1: Psycho-education Tool

* Objective: Develop and evaluate a tool to support healthcare providers and patients in understanding and addressing sexual and domestic violence, trauma, and their impacts on well-being.
* Tool Description: A set of cards presented in a calendar format, featuring illustrations on one side and explanatory text on the other.

Target Groups: Healthcare providers and victims/patients.

* Development process: The tool was developed based on literature and input from experts and stakeholders during regular meetings.
* Testing Phase: The tool will undergo a pilot study in selected hospitals and non-profit organizations (NGOs) working with victims of violence.
* Evaluation: The tool's acceptability, usability, and relevance to the recovery process will be assessed through feedback collected via questionnaires from both healthcare providers and victims/patients.

Sub-Study 2: Guidelines Older Adults

* Objective: Develop and implement guidelines for screening violence among older adults and providing appropriate care for victims of various forms of violence (psychological, physical, (socio-)economic, and sexual).
* Tool Description: A guideline that includes a screening protocol, care and referral pathways, and theoretical background on the topic.
* Target Group: Older adults with sufficient cognitive abilities.
* Development Process: The guidelines are informed by a literature review, expert, and stakeholder input through regular meetings and focus groups, and a pilot study involving cognitively capable older adults in the geriatric departments of four hospitals.
* Testing Phase: The screening protocol is integrated into standard care procedures, such as intake interviews or geriatric assessments. It is implemented by multidisciplinary professionals, including physicians, nurses, psychologists, occupational therapists, and social workers.
* Evaluation: Feedback on the guidelines is collected from healthcare providers via questionnaires. Older adults themselves are not directly involved in the evaluation, as the screening protocol is intentionally embedded discreetly within standard care procedures.

Training and Support The project includes a robust training component delivered through educational online modules designed to equip healthcare providers with the knowledge and skills necessary to effectively use the tools and guidelines developed.

Languages and Application The study materials and procedures are conducted in both French and Dutch, reflecting Belgium's bilingual context.

Significance This project highlights the importance of tailored support for victims of violence and a systematic approach to care within clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Substudy 1: Psycho-education Tool

* Healthcare Providers: In-hospital healthcare providers who used the psycho-education tool during the pilot phase with a victim of violence.
* Victims/Patients: Victims of violence aged 16 years or older who received psycho-education from an in-hospital healthcare provider during the pilot phase.

Substudy 2: Guideline

* Healthcare Providers: In-hospital healthcare providers who used the guideline during the pilot phase with an older adult.
* Older Adults/Patients: Older adults with sufficient cognitive abilities who were admitted to the geriatric department (either for a day clinic or a longer stay).

Exclusion Criteria:

Substudy 1: Psycho-education tool

* Victims under the age of 16. Substudy 2: Guideline
* Older adults with cognitive impairments.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Enhanced identification, care, and referral processes for victims of violence. | Conducting the psycho-education tool or guideline will not take more than 30 minutes in total.
  Conduct a pilot study to evaluate a recently developed psycho-education tool and guideline for healthcare providers (Operation Alert study). These tools aim to enhance the delivery of psycho-education to victims of violence and improve the identification of and care for older victims of violence. The tools are evaluated through a self-developed questionnaire based on the theoretical framework of acceptability by Sekhon (2022), assessing 7 constructs: affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.
  In substudy 1, healthcare providers complete 11 open-ended questions and demographics, while patients answer 9 closed questions (Likert 1-5) and 10 open-ended ones. In substudy 2, healthcare providers piloting the guideline have to complete 6 open questions, 11 closed questions (Likert 1-5), and demographics. There are also 11 open-ended questions with no obligation to complete.

SECONDARY OUTCOMES:
Evaluating the feasibility and acceptability of the psycho-education tool and guideline in clinical practice. | An evaluation is completed after testing the psycho-education tool or guideline and takes approximately 10 minutes.
  Targeted adjustments and finalization of the psycho-education tool and guidelines can be made based on the feedback obtained from questionnaires of healthcare providers (substudy 1 and 2) and patients/victims (substudy 1).
  The tools are evaluated by using a self-developed questionnaire based on the theoretical framework of acceptability (TFA) by Sekhon (2022). The questions comprise seven component constructs: affective attitude, burden, ethicality intervention coherence, opportunity costs, perceived effectiveness and self-efficacy.
  The framework presents a generic TFA questionnaire to evaluate the acceptability of interventions from the perspectives of recipients. It can be adapted to assess acceptability of any healthcare intervention. Its development was guided by theory, previous research, and stakeholder input.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Keygnaert, Ph.D, Principal Investigator — Ghent University Hospital and Ghent University (VIORESC)
Locations (10):
- Belgium (10):
  - Aditi ASBL/vzw, Antwerp
  - Vertrouwenscentrum Kindermishandeling Antwerpen, Antwerp
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Vertrouwenscentrum Kindermishandeling Brussel, Brussels
  - SOSEnfants Bruxelles ASBL, Brussels
  - SOSEnfants Charleroi ASBL, Charleroi
  - Ghent University Hospital, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
  - AZ Delta, Roeselare
  - SOSEnfants Namur ASBL, Saint-Servais

IPD SHARING:
Plan to Share IPD: No
Individual patient data are anonymized and encrypted to ensure privacy and security. The research specifically addresses violence, with a focus on sexual and domestic violence among participants aged 16 and older. Sharing any individual patient data would breach the confidentiality of this sensitive group and violate European GDPR regulations.

REFERENCES:
- [Derived] Boven C, Nobels A, Berg N, Van Den Noortgate N, Courtens N, Keygnaert I. Screening and Caring for Older Adults Affected by Sexual or Other Types of Violence: A Pilot Study at Three Belgian Geriatric Departments. Healthcare (Basel). 2025 Dec 20;14(1):16. doi: 10.3390/healthcare14010016. PMID 41516947
- See also: Related Info — https://operatiealert.be/
- See also: Related Info — https://operationalerte.be/